CLINICAL TRIAL: NCT04064944
Title: Comparison of the Efficacy and Safety of Immunoadsorption and Plasma Exchange for Acute Attack of Refractory Neuromyelitis Optica Spectrum Disorders: a Prospective, Multicenter, Single-blind, Randomized Controlled Clinical Trial
Brief Title: Comparison of the Efficacy and Safety of Immunoadsorption and Plasma Exchange for Acute Attack of Refractory Neuromyelitis Optica Spectrum Disorders
Acronym: CAMPUS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other); Guangdong 999 Brain Hospital (Other)
Responsible Party: Principal Investigator, Wei Qiu, professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20190705
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: Neuromyelitis Optica Spectrum Disorder; immunoadsorption; plasma exchange; acute attack; refractory
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunoadsorption group (Experimental): patients' blood purification treatment protocal is Protain A Immunoadsorption method.
  Interventions: Device: blood purification equipment
- Plasma exchange group (Experimental): patients' blood purification treatment protocal is Plasma exchange method.
  Interventions: Device: blood purification equipment

INTERVENTIONS:
Device: blood purification equipment — The subjects enrolled in this study will undergo blood purification treatment, and will be randomized into either immunoadsorption group or plasma exchange group, and the following indicators will be evaluated: (1) changes in EDSS scores and visual acuity before and after treatment; (2) changes in AQP4-IgG levels; (3) the safety of immunoadsorption treatment.

SUMMARY:
Neuromyelitis optica spectrum disorder (NMOSD) is one common demyelinating disease of the central nervous system in young adults, with high rate of disability and recurrence, and poor natural course, which can cause a serious burden on families and society. To today, there is still a lack of prospective, multi-center, large sample clinical trial evidence for the treatment and prognosis of acute attack of NMOSD patients. This study will conduct a prospective, multi-center, single-blind, randomized controlled clinical trial of acute attacked NMOSD patients in China. The researchers plan to collect 144 NMOSD patients with acute attack in three research centers of Guangzhou (the Third Affiliated Hospital of Sun Yat-sen University, the Zhongshan Ophthalmic Center of Sun Yat-sen University, and the Guangdong 999 Brain hospital), to study the safety and efficacy of immunoadsorption therapy.

The subjects will be randomized into immunoadsorption group and plasma exchange group, and the following indicators will be evaluated: (1) changes in EDSS scores and visual acuity before and after treatment; (2) changes in AQP4-IgG levels; (3) the safety of immunoadsorption treatment.

This study is aimed to determine the efficacy and safety of immunoadsorption therapy for acute attack of refractory NMOSD patients, and to provide more sufficient clinical evidence for the therapy selection for acute phase of NMOSD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should meet the 2015 International NMOSD with acute attacks diagnostic criteria (including first episodes and recurrences)
2. When NMOSD Patients with acute attacks undergo a course of hormone shock therapy (5-10g total methylprednisolone), EDSS ≥ 6.0 or visual acuity ≤ 20/200
3. Serum AQP4-IgG positive (CBA test)

Exclusion Criteria:

1. Weight <25Kg
2. Nursing or pregnant women
3. Unable to establish a peripheral or central vascular access
4. The use of rituximab and gamma-ball shocks within 3 months prior to enrollment
5. Using immunoadsorption and/or plasma exchange therapy within 3 months before enrollment
6. ACEI drugs must be taken within 1 week before the first treatment and during treatment and cannot be stopped

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in EDSS scores | 4 weeks after the last treatment vs.baseline ( first treatment)
  Changes in EDSS scores of 4 weeks after the last treatment of plasma exchange or immunoadsorption compared with the first treatment

SECONDARY OUTCOMES:
Comparison of follow-up results of EDSS scores | the next 1 day, 1 week, 2 weeks, 3 months after the last treatment vs. baseline (that of the time before first treatment)
  Comparation of the changes in EDSS scores of the next day, 1 week, 2 weeks, 3 months after the last plasmapheresis or immunoadsorption treatment vs. that before the first treatment
Comparison of follow-up results of LogMAR | the next 1 day, 1 week, 2 weeks, 3 months after the last treatment vs. baseline (that of the time before first treatment)
  Comparation of the changes in LogMAR of the next day, 1 week, 2 weeks, 3 months after the last plasmapheresis or immunoadsorption treatment vs. that before the first treatment (NMO patients)
Comparison of follow-up results of AQP4-IgG level | the next 1 day, 1 week, 2 weeks, 3 months after the last treatment vs. baseline (that of the time before first treatment)
  Comparation of the changes in AQP4-IgG level of the next day, 1 week, 2 weeks, 3 months after the last plasmapheresis or immunoadsorption treatment vs. that before the first treatment

IPD SHARING:
Plan to Share IPD: No